CLINICAL TRIAL: NCT03875157
Title: To Evaluate the Safety, Tolerability, and Initial Efficacy of IBI318 in Patients With Advanced Malignancy, Multicenter, IA/IB Study
Brief Title: Study of IBI318 in Participants With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI318A101
Record Dates: First submitted 2019-02-28; First posted 2019-03-14 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Advanced Malignancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- IBI318 DL1 (Experimental)
  Interventions: Biological: IBI318
- IBI318 DL2 (Experimental)
  Interventions: Biological: IBI318
- IBI318 DL3 (Experimental)
  Interventions: Biological: IBI318
- IBI318 DL4 (Experimental)
  Interventions: Biological: IBI318
- IBI318 DL5 (Experimental)
  Interventions: Biological: IBI318
- IBI318 DL6 (Experimental)
  Interventions: Biological: IBI318
- IBI318 DL7 (Experimental)
  Interventions: Biological: IBI318
- IBI318 DL8 (Experimental)
  Interventions: Biological: IBI318
- IBI318 DL7b (Experimental)
  Interventions: Biological: IBI318
- IBI318 DL8b (Experimental)
  Interventions: Biological: IBI318
- IBI318 RP2D (Experimental)
  Interventions: Biological: IBI318

INTERVENTIONS:
Biological: IBI318 — 0.3 mg intravenous infusion, C1D1 and afterwards Q2W
  Arms: IBI318 DL1
Biological: IBI318 — 1 mg intravenous infusion, C1D1 and afterwards Q2W
  Arms: IBI318 DL2
Biological: IBI318 — 3 mg intravenous infusion, C1D1 and afterwards Q2W
  Arms: IBI318 DL3
Biological: IBI318 — 10 mg intravenous infusion, C1D1 and afterwards Q2W
  Arms: IBI318 DL4
Biological: IBI318 — 30 mg intravenous infusion, C1D1 and afterwards Q2W
  Arms: IBI318 DL5
Biological: IBI318 — 100 mg intravenous infusion, C1D1 and afterwards Q2W
  Arms: IBI318 DL6
Biological: IBI318 — 300 mg intravenous infusion, C1D1 and afterwards Q2W
  Arms: IBI318 DL7
Biological: IBI318 — 600 mg intravenous infusion, C1D1 and afterwards Q2W
  Arms: IBI318 DL8
Biological: IBI318 — Intravenous infusion, C1D1 and afterwards Q3W
  Arms: IBI318 DL7b
Biological: IBI318 — Intravenous infusion, C1D1 and afterwards Q3W
  Arms: IBI318 DL8b
Biological: IBI318 — Intravenous infusion Q3W
  Arms: IBI318 RP2D

SUMMARY:
An open label, multicenter, phase Ia/Ib study to evaluate the safety, tolerability, and initial efficacy of IBI318 in the treatment of patients with advanced malignancies.

DETAILED DESCRIPTION:
An open label, multicenter, phase Ia/Ib study to evaluate the safety, tolerability, and initial efficacy of IBI318 in the treatment of patients with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form
2. Men or women 18 years or older
3. Expected survival time ≥ 12 weeks
4. Tumor assessment according to RECIST v1.1, at least one measurable lesion
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Have adequate organ and bone marrow function
7. Male participants and female participants must agree to use contraception during the treatment period and within 180 days after the treatment period
8. Female subjects must not be pregnant or breastfeeding. If premenopausal, negative urine or serum pregnancy tests are required
9. Ia: Subjects with locally advanced, recurrent or metastatic histologically or cytologically confirmed solid tumors or hematologic tumors and are refractory or intolerant to existing standard treatments
10. Ib: Metastatic non-small cell lung cancer, advanced liver cancer, advanced esophageal squamous cell cancer, advanced gastric cancer, or other tumors that have been proved by histology or cytology with initial therapeutic effect in Phase Ia

Exclusion Criteria:

1. Previous exposure to immunotherapy including but not limited to, anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies, excluding therapeutic anti-tumor vaccine
2. Participation in another interventional clinical study, an observational (non-interventional) clinical study, or a follow-up phase of an interventional study
3. Receive last anti-tumor treatment within 4 weeks prior to the first dose of study drug
4. Use of immunosuppressive drugs within 4 weeks prior to the first dose of study drug
5. Require long-term steroid therapy or any other form of immunosuppressive therapy not including inhaled steroids
6. Toxicity (excluding hair loss or fatigue) caused by previous antitumor therapy that did not recover to NCI CTCAE v 5.0 level 0-1 within 4 weeks prior to the first dose of study drug
7. Received major surgery or has unhealed wounds, ulcers, or fractures within 4 weeks prior to the first dose of study drug
8. Expect to receive other anti-tumor treatments during study (allowing palliative radiotherapy)
9. History of infectious pneumonitis that required steroids or has current pneumonitis
10. Known active untreated CNS metastases and/or spinal cord compression and/or cancerous meningitis, or with a history of soft meningeal cancer
11. Active autoimmune disease that has required systemic treatment in past 2 years
12. Known active Hepatitis B or Hepatitis C virus
13. Uncontrolled concomitant diseases or neurological, psychiatric/social conditions that could affect study compliance, significantly increase the risk of adverse events, or affect the participant's ability to provide written informed consent
14. Known history of human immunodeficiency virus (HIV) infection
15. Known history of active tuberculosis (TB) or active syphilis
16. History of allogeneic organ transplantation or hematopoietic stem cell transplantation
17. Accompanied by uncontrolled third interstitial fluids requiring repeated drainage, such as pleural effusion, ascites, pericardial effusion, etc.
18. Known severe allergic reactions to other monoclonal antibodies or are allergic to any IBI318 formulation component
19. Female subjects who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing dose-limiting toxicities (DLTs) | 28 days within first dose in phase Ia
Number of participants experiencing clinical and laboratory adverse events (AEs) | Up to 90 days post last dose
Number of all study participants who demonstrate a tumor response | up to 24 months

SECONDARY OUTCOMES:
The area under the curve (AUC) of plasma concentration of drug against time after administration of IBI318 | Up to 90 days post last dose
Maximum concentration (Cmax) after first dose interval of IBI318 | Up to 90 days post last dose
Time at which maximum concentration (Tmax) occurs for IBI318 | Up to 90 days post last dose
The half-life (t1/2) of IBI318 in plasma | Up to 90 days post last dose
Positive rate of ADA and Nab | Up to 90 days post last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China